CLINICAL TRIAL: NCT04022590
Title: Tri-service General Hospital
Brief Title: Cardiopulmonary Training in the Victims With Multiple Morbidities by Application of Novel Heart Rate Sensing Clothes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shang-Lin Chiang (Other)
Responsible Party: Sponsor-Investigator, Shang-Lin Chiang, Attending physician, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Smart clothes
Record Dates: First submitted 2019-05-18; First posted 2019-07-17 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Degeneration Muscle; Multiple Morbidities; Heart; Complications

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-clothes (Experimental): The participants with E-clothes do aerobic training at home
  Interventions: Device: E-clothes; Behavioral: Healthy consultation
- Home exercise (Active Comparator): The participants with healthy consultation do aerobic training at home.
  Interventions: Behavioral: Healthy consultation

INTERVENTIONS:
Device: E-clothes — The E-clothes could prove heart rate or heart rate variability(HRV) information to the participants' smart phone by blue tooth. Then the smart phone will calculate and provide the suitable aerobic training intensity by the microphone when the participants do aerobic training.
  Arms: E-clothes
Behavioral: Healthy consultation — Healthy consultation will educate the participants do aerobic training three times a week for 3 months. And the each training period is at least 30 minutes.

SUMMARY:
Investigators assume that the wearable clothes can be applied to home-based health care and integrated into a case management model through telehealthcare. While prior to complete the case management, the feasibility should be tested and evaluate its reliability and validity of the physical information collected from the clothes. Therefore, investigators try to conduct a feasibility study to evaluate the reliability and validity of the exercise heart rate sensing e-clothes and after that, investigators will incorporate this wearable clothes to home-based exercise training as one of the major components in our case management model.

DETAILED DESCRIPTION:
Easy-to-use and service touch points allow patients/ users to realize the value and status of their physiological functions/ parameters based on their evidence is important. According to the U.S. survey, 90% of people can change their lifestyle behaviors, improve their personal health awareness, achieve holistic health care and improve their quality of life due to "Quantify Self". Therefore, a broader health care system, health consumption services or ecological system has been building to integrate health care resources, extend health care services from hospital to communities and individual' homes. When people consume in their daily life, immediate public health guidance or professional intervention can be offered at the same time, not only can effectively maintain individuals' health, early detection of possible physiological signs/ parameters, can also delay the progression of the disease and reduce the burden of first-line health care workers. Therefore, it is the era of smart healthcare that provides a health service platform with APPs(Applications) to provide personalized integrated medical services. However, in order to monitor or evaluate the effect of treatment (i.e., exercise training) still needs to be provided through the actual feedback of individual physiological data.

Clothes with smart function which is able to connect with social media and APPs has been promoting and marketing as smart sports or lifestyle-monitor goods, such as exercise-related physical parameters and sleep quality quantifying. Sleep physiology information collected through the clothes including degree and quality of sleep can be recorded and transmitted to the remote health system via APP and cloud service platform. On this cloud platform, health information can exchange with clinician's physicians, offering advises for users to whether to go to the hospital for further examination.

ELIGIBILITY:
Inclusion Criteria:

* more than two chronic disease.(multiple morbidity)
* able to speak and understand Mandarin
* able to walk without assistance
* able to use smart phones and understand how to use the e-clothes and related app
* agreed to be randomized to one of the two groups

Exclusion Criteria:

* a history of cancer
* confirmed psychiatric disease
* inability to participate due to comorbid neurological and musculoskeletal conditions
* a history of arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity (VO2 max in ml/kg/min ) | 30 minutes
  Maximal VO2 during testing, also means aerobic capacity
Working load in watt | 30 minutes
  Maximal Working load during testing
Rest/Max Heart rate in beat/min | 30 minutes
  resting and maximal heart rate during exercise testing,
O2 pulse in ml/beat, | 30 minutes
  It means the heart pumps O2 volume by each heart beat, and also means left ventricle function.
systolic and diastolic blood pressure in mm Hg, | 30 minutes
  The resting and maximal blood pressure during exercise testing

SECONDARY OUTCOMES:
Physical activity (scores) | 10 minutes
  The participants' weekly physical activity will be assessed by a research nurse using the International Physical Activity Questionnaire (IPAQ)-short form, Chinese version, which has well-established reliability and validity (Liou, Jwo, Yao, Chiang, & Huang, 2008). This 7-item instrument measures time (minute) of physical activity including housework, transportation, leisure activity, and moderate-to-vigorous-intensity physical activity for the past 7 days.

OTHER OUTCOMES:
Quality of life (scores) | 20 minutes
  The indicator of quality of life in this study will use Short-Form 36 to evaluate. The Taiwan standard version SF-36 developed through the collaboration of Drs. Jui-Fen Rachel Lu et al. in 1996 showed well-established reliability and validity.
Depression (scores) | 10 minnutes
  Symptoms of depression will be assessed using the 21-item BDI, which is a self-report questionnaire frequently used to examine depressive level during the previous two weeks (Beck, Steer, & Brown, 1996)

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No